CLINICAL TRIAL: NCT01853449
Title: Effects of Inhaled Fentanyl Citrate on Perceived Respiratory Discomfort (Dyspnea) During Exercise in the Presence of External Thoracic Restriction
Brief Title: Inhaled Fentanyl Citrate & Dyspnea
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dennis Jensen, Ph.D., Assistant Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A02-M16-13B Fentanyl
Record Dates: First submitted 2013-05-07; First posted 2013-05-15 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Dyspnea
Keywords: Fentanyl Citrate; Opioids; Exercise
MeSH Terms: conditions — Dyspnea; Motor Activity | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CWS+Fentanyl Citrate (250 mcg) (Experimental): Chest wall strapping to reduce vital capacity by 20% of its baseline value + single-dose inhalation of nebulized fentanyl citrate (250 mcg)
  Interventions: Drug: Fentanyl Citrate; Other: CWS
- CWS+0.9% saline placebo (Placebo Comparator): Chest wall strapping to reduce vital capacity by 20% of its baseline value + single-dose inhalation of 0.9% saline placebo
  Interventions: Other: CWS; Drug: Placebo
- No CWS+Fentanyl Citrate (250 mcg) (Active Comparator): No chest wall strapping (unloaded control) + single-dose inhalation of nebulized fentanyl citrate (250 mcg)
  Interventions: Drug: Fentanyl Citrate
- No CWS+0.9% saline placebo (Placebo Comparator): No chest wall strapping (unloaded control) + single-dose inhalation of 0.9% saline placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fentanyl Citrate
  Arms: CWS+Fentanyl Citrate (250 mcg); No CWS+Fentanyl Citrate (250 mcg)
Other: CWS — Chest wall strapping to reduce vital capacity by 20% of its baseline value
  Other Names: chest wall strapping
  Arms: CWS+0.9% saline placebo; CWS+Fentanyl Citrate (250 mcg)
Drug: Placebo — 0.9% saline
  Arms: CWS+0.9% saline placebo; No CWS+0.9% saline placebo

SUMMARY:
"Dyspnea" refers to the awareness of breathing discomfort that is typically experienced during exercise in health and disease. In various participant populations, dyspnea is a predictor of disability and death; and contributes to exercise intolerance and an adverse health-related quality-of-life. It follows that alleviating dyspnea and improving exercise tolerance are among the principal goals of disease management. Nevertheless, the effective management of dyspnea and activity-limitation remains an elusive goal for many healthcare providers and current strategies aimed at reversing the underlying chronic disease are only partially successful in this regard. Thus, research aimed at identifying dyspnea-specific medications to complement existing therapies for the management of exertional symptoms is timely and clinically relevant. The purpose of this study is to test the hypothesis that single-dose inhalation of fentanyl citrate (a mu-opioid receptor antagonist) will improve the perception of dyspnea during strenuous exercise in healthy, young men in the presence of an external thoracic restriction. To this end, the investigators plan compare the effects of inhaled 0.9% saline placebo and inhaled fentanyl citrate (250 mcg) on detailed assessments of neural respiratory drive (diaphragm EMG), ventilation, breathing pattern, dynamic operating lung volumes, contractile respiratory muscle function, cardio-metabolic function and dyspnea (sensory intensity and affective responses) during symptom-limited, high-intensity, constant-work-rate cycle exercise testing with and without external thoracic restriction in healthy, men aged 20-40 years.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 20-40 years
* FEV1 ≥80% predicted
* FEV1/FVC >70%

Exclusion Criteria:

* Current or ex-smoker
* Body Mass Index <18.5 or >30 kg/m2
* History of cardiovascular, vascular, respiratory, renal, liver, musculoskeletal, endocrine, neuromuscular and/or metabolic disease/dysfunction
* Taking doctor prescribed medications
* History of using pain-relieving (opioid) and/or anti-depressant medications in the previous 6 weeks
* Allergy to latex
* Allergy to lidocaine or its "caine" derivatives

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sensory intensity (Borg 0-10 scale) ratings of dyspnea at isotime | Participants will be followed until all study visits are completed, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, Ph.D., Principal Investigator — McGill University
Locations (1):
- Montreal Chest Institute; McGill University Health Center & McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kotrach HG, Bourbeau J, Jensen D. Does nebulized fentanyl relieve dyspnea during exercise in healthy man? J Appl Physiol (1985). 2015 Jun 1;118(11):1406-14. doi: 10.1152/japplphysiol.01091.2014. Epub 2015 Mar 12. PMID 26031762
- See also: Clinical Exercise & Respiratory Physiology Laboratory (CERPL) of McGill University — http://www.mcgill.ca/cerpl